CLINICAL TRIAL: NCT05291286
Title: A Pilot Proof of Concept Pharmacokinetic/Pharmacodynamic Study of BXQ-350 in Cancer Patients Exposed to Oxaliplatin and/or Taxane-Based Chemotherapy
Brief Title: BXQ-350 Pharmacokinetic/Pharmacodynamic Study in Cancer Patients
Acronym: RETRO
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Bexion Pharmaceuticals, Inc. (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: BXQ-350.AH
Record Dates: First submitted 2022-03-11; First posted 2022-03-22 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Neuropathy;Peripheral; Chemotherapy-induced Peripheral Neuropathy
MeSH Terms: conditions — Neuritis

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to 1 of 2 treatment arms (BXQ-350 or placebo) in a 1:1 ratio for the first two treatment cycles. At the end of the second treatment cycle, participants will be unblinded to their individual treatment assignment. Participants who received placebo will be offered 2 cycles of open-label BXQ-350. Participants who received BXQ-350 in Cycles 1 and 2 will continue to the Post-Treatment Follow-Up. If placebo participants elect to forego BXQ-350 at the time of unblinding, their participation in the study will end following an end of study visit.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: randomized, placebo controlled, double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BXQ-350 (Experimental): BXQ-350 will be administered by IV infusion
  Interventions: Drug: BXQ-350
- Placebo (Placebo Comparator): Placebo (0.9% normal saline) will be administered by IV infusion
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BXQ-350 — BXQ-350 is a novel anti-neoplastic therapeutic agent configured from two components: Saposin C (SapC), an expressed (human) lysosomal protein, and the phospholipid dioleoylphosphatidyl-serine (DOPS), a phospholipid located on cell membranes (clinical formulation BXQ-350). BXQ-350 will be administered by intravenous (IV) infusion
  Other Names: SapC-DOPS
  Arms: BXQ-350
Other: Placebo — Placebo will be 0.9% normal saline of matching volume to BXQ-350 administered by intravenous (IV) infusion
  Arms: Placebo

SUMMARY:
This study will assess pharmacokinetic (PK)/pharmacodynamic (PD) relationships and whether BXQ-350 may decrease the intensity and/or duration of chemotherapy induced peripheral neuropathy (CIPN) thereby improving quality of life (QoL) in cancer patients who have been exposed to oxaliplatin and/or taxane-based chemotherapy. This study includes two randomized, placebo controlled, blinded treatment cycles of BXQ-350/placebo, an optional open-label BXQ-350 treatment period, and an unblinded Post-Treatment Follow-up period.

DETAILED DESCRIPTION:
BXQ-350 is a novel anti-neoplastic therapeutic agent configured from two components: Saposin C (SapC), an expressed (human) lysosomal protein, and the phospholipid dioleoylphosphatidyl-serine (DOPS), a cell membrane phospholipid (clinical formulation BXQ-350).Due to the presumed mechanism of action of BXQ-350, Bexion anticipates that it may have an impact on ceramides, sphingosine-1-phosphate (S1P), and inflammatory cytokine levels. In addition, pre-clinical results demonstrated that BXQ-350 induced neurite generation and protection in vitro in the PC-12 and NS20Y cell lines and significantly decreased oxaliplatin-induced cold allodynia in a model of CIPN. Thus BXQ-350 may represent a new approach to deliver a neuropathy benefit.

The unique combination of SapC-DOPS along with its proven safety profile and possible neuropathy benefit makes BXQ-350 a worthwhile candidate to test on cancer patients affected by CIPN. The aim of this pilot proof-of-concept study is to assess PK/PD relationships in cancer patients with CIPN symptoms in order to determine the impact BXQ-350 has on ceramide, S1P, and inflammatory cytokine levels; thereby potentially reducing the intensity and/or duration of CIPN, improving QoL, and establishing these signaling molecules as biomarkers in future studies.

This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.)

ELIGIBILITY:
Inclusion Criteria:

Participants who meet the following criteria will be considered eligible to participate in the clinical study:

1. Age ≥ 18 years of age at the time of signing the informed consent.
2. Have a diagnosis of cancer.
3. Have symptoms of CIPN persisting ≥6 months and determined by the participant's treating physician to be caused by prior exposure to oxaliplatin or taxane-based chemotherapy.
4. Have an EORTC QLQ-CIPN20 score of 3 (quite a bit) or 4 (very much) on at least 1 of the 6 questions pertaining to numbness, tingling, or pain in the fingers/hands or toes/feet.
5. Have a life expectancy > 12 months.
6. Have ECOG Performance Status of 0 or 1.
7. Have acceptable liver function defined as:

   * Total serum bilirubin ≤ 1.5 x upper limit of normal (ULN) for the study site. In participants with known Gilbert Syndrome, total bilirubin ≤ 3 x ULN, with direct bilirubin ≤ 1.5 x ULN).
   * Aspartate transaminase (AST), serum glutamic oxaloacetic transaminase (SGOT), alanine transaminase (ALT), serum glutamic pyruvic transaminase (SGPT) ≤ 3 x ULN (if liver metastases are present, then ≤ 5 x ULN is allowed).
   * Serum albumin ≥ 3 g/ dL.
8. Have acceptable renal function defined as:

   * Creatinine clearance ≥ 50 mL/minute calculated using the Cockcroft-Gault formula (Cockcroft 1976):

   CCr = {((140 - age) x weight kg) / (72 x SCr)} x 0.85 (if female).
   * Urine dipstick protein ≤ 1 + (30 - 70 mg/dL) OR urine protein/creatinine ratio of ≤ 1, OR 24 hour urine protein < 1g/24 hours.
9. Have acceptable bone marrow function defined as:

   * White blood cell count > 3,000 cells / mm3 OR absolute neutrophil count ≥ 1,500 cells / mm3.
   * Platelet count ≥ 100,000 cells / mm3 (unsupported, no transfusion within 7 days of enrollment).
   * Hemoglobin > 9.0 g/dL (unsupported, no transfusion within 7 days of enrollment).
10. Have acceptable coagulation parameters (anti-coagulation allowed) defined as:

    * International normalized ratio ≤ 2 x ULN unless on anticoagulation or prothrombin time within normal limits.
    * Activated partial thromboplastin time within normal limits.
11. Have a negative serum pregnancy test result at screening (females of childbearing potential [FCBP] only). Not applicable to participants who are surgically sterile (i.e., bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy) or who are post menopausal. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.
12. Contraceptive use by men and women must be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. FCBP whose partner(s) are non-sterilized male participants whose sexual partner(s) are FCBP must abstain from heterosexual activity or agree to use an acceptable method of contraception according to the followingguidelines:

    * The reliability of sexual abstinence for male and/or female enrollment eligibility needs to be evaluated in relation to the duration of the entire period of risk associated with study interventions and the preferred and usual lifestyle of the participant. Total sexual abstinence is an acceptable method provided it is the usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post ovulation methods), the rhythm method, and withdrawal are not acceptable methods of contraception.
    * Non-sterilized Male Participants:

      * Must use an acceptable method of contraception such as male condom plus spermicide during the entire period of risk associated with study interventions which includes the total duration of the study and the drug washout period (6 months after the last dose of study intervention) and refrain from sperm donation or banking throughout this period.
      * Vasectomized males are considered fertile and should still use a male condom plus spermicide as indicated above.
      * Even if the female partner is pregnant, male participants should still use a condom plus spermicide, as indicated above.
      * Female partners (of childbearing potential) of male participants must also use a highly effective method of contraception during the entire period of risk associated with study interventions as described above.
    * FCBP

      * Must use a highly effective method of contraception and avoid breastfeeding during the entire period of risk associated with study interventions which includes the total duration of the study and the drug washout period (9 months after the last dose of study intervention) and have been stable on their chosen method of birth control for a minimum of 3 months before entering the study.
      * Non-sterilized male partners must also use a male condom plus spermicide during the entire period of risk associated with study interventions as described above.
    * A highly effective method of contraception is defined as one that results in a low failure rate (less than 1% per year) when used consistently and correctly. Note that some contraception methods are not considered highly effective.

    The participants chosen method(s) must be confirmed as highly effective prior to study entry.
13. Participant is capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

Participants must not meet any of the following criteria:

1. Have received chemotherapy known to cause CIPN in the last 12 months.
2. Currently receiving or expected to initiate chemotherapy for the treatment of an active cancer during the study period; cancer therapies utilized to maintain remission that are not known to cause or exacerbate peripheral neuropathy, as well as maintenance endocrine/hormonal/immune therapy for cancer are allowed. Continuation of polyadenosine diphosphate-ribose polymerase (PARP) inhibitors or other targeted therapies not associated with peripheral neuropathy is permitted.
3. Have Type 1 or 2 diabetes mellitus.
4. Have a family history of a genetic/familial neuropathy.
5. Have pre-existing clinical neuropathy ≥ Grade 2 per CTCAE v5.0 from any cause.
6. Currently taking daily oral steroids exceeding prednisone 10 mg daily or its equivalent.
7. Participants with brain metastases may participate provided they are clinically stable for at least 4 weeks prior to study entry, have no evidence of new or enlarging metastases and are off steroids for at least 7 days.
8. Have had major surgery within 28 days prior to randomization or have not recovered from major side effects of the surgery if more than 4 weeks have elapsed since surgery. Minor outpatient procedures are allowed.
9. Have poorly controlled hypertension defined as blood pressure > 150/90 mmHg on at least 2 repeated determinations prior to screening or on day of screening.
10. Have a history of cardiac dysfunction including:

    * Myocardial infarction within 6 months prior to initiation of screening.
    * History of documented congestive heart failure (New York Heart Association functional classification III-IV) within 6 months prior to initiation of screening.
    * Active cardiomyopathy.
    * Electrocardiogram with QTc > 470 milliseconds at screening.
11. Have uncontrolled severe infections (acute or chronic) including HIV, Hepatitis B or C.
12. Have active poor wound healing (delayed healing, wound infection or fistula).
13. Have evidence of active clinically significant bleed (e.g., gastrointestinal bleed, hemoptysis, or gross hematuria) at screening.
14. Are breast feeding or pregnant, confirmed by a positive serum human chorionic gonadotropin (hCG) laboratory test.
15. Have other concurrent severe and/or uncontrolled medical condition that would, in the Investigator's judgment contraindicate the participant's participation in the clinical study or obscure proper assessment of safety and toxicity of the prescribed regimen.
16. Received prior treatment with any investigational drug within 4 weeks (28 + 3 days) prior to randomization.
17. Are receiving any agent for the treatment, prevention, or with known/hypothesized efficacy for peripheral neuropathy and have had the dose adjusted within 28 days prior to BXQ-350/placebo dosing. Agents include but not limited to: narcotics, gabapentin, pregabalin, venlafaxine, duloxetine, amitriptyline, nortriptyline, topiramate, lamotrigine, or anti- neuropathic pain topical cream.

    * Note: Participants who have been on a stable dose of an above agent (or agents) for at least 28 days prior to BXQ-350/placebo dosing are eligible and may continue receiving the agent during the study. Participants may continue taking acetaminophen for neuropathy pain during the study.
18. Have a known sensitivity to any component of BXQ-350 (SapC and DOPS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 6 months
  To evaluate the Cmax of BXQ-350.
Ceramide | 6 months
  To evaluate ceramide levels following administration of BXQ-350.
S1P levels | 6 months
  To evaluate S1P levels following administration of BXQ-350.
Cytokine levels | 6 months
  To evaluate cytokine levels following administration of BXQ-350.
Quality of Life (QoL) | 6 months
  To evaluate QoL in patients with neuropathy receiving BXQ-350. QoL will be measured utilizing the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30).
Total Sensory Neuropathy | 6 months
  To evaluate neuropathy symptoms in patients with neuropathy receiving BXQ-350. Total sensory neuropathy scores will be obtained from the EORTC QLQ-CIPN20 questionnaire.
CIPN Assessment | 6 months
  To evaluate CIPN symptoms in patients with neuropathy receiving BXQ-350 utilizing the CIPN Assessment Tool questionnaire.

SECONDARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events as Assessed by CTCAE v5.0 | 6 months
  To further assess the overall safety and tolerability of BXQ-350as evidenced by the incidence of treatment emergent adverse events assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - CTI Clinical Research Center, Cincinnati, Ohio
  - The Ohio State Unviersity, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No